CLINICAL TRIAL: NCT01024764
Title: Observational Study of the Phase I Safety and Immunogenicity Trial of Recombinant HIV-1 Tat in HIV-1 Uninfected Adult Volunteers
Brief Title: Observational Study of the Preventive Trial With HIV-1 Tat Protein
Acronym: ISS OBS P-001
Status: Completed | Type: Observational
Sponsor: Istituto Superiore di Sanità (Other)
Responsible Party: Barbara Ensoli, CNAIDS - Istituto Superiore di Sanita
Other Study IDs: ISS OBS P-001
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2010-02

CONDITIONS: Healthy Subjects
Keywords: HIV; Tat protein; Preventive vaccine

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, serum, PBMCs
Oversight: Data Monitoring Committee: No

SUMMARY:
The results of the Phase I Safety and Immunogenicity Trial of Recombinant HIV-1 Tat (ISS P-001 and ISS T-001) indicate that the vaccine based on the recombinant Tat protein is safe, well tolerated and immunogenic. The present study is intended to extend the follow-up of the volunteers for additional 3 years to evaluate the persistence of the anti-Tat humoral and cellular immune response. The results of the present study will be key for the design of future phase II trials, particularly for the definition of the optimal schedule for boosting immunizations.

All individuals (20) will be enrolled in a 120-weeks observational study and monitored every 24 weeks for the following 3 years. During these visits, in addition to the hematological and biochemical assessment, the anti-Tat specific humoral and cellular immune responses will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Previous participation to the Phase I Clinical Trial ISS P-001

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Subjects previously included in the Preventive Phase I Clinical Trial with Tat protein
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2007-11; Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the persistence of specific immune responses, volunteers will be monitored for anti-Tat specific antibodies, anti-Tat proliferative response and in vitro γIFN and IL-4 production in response to Tat (Elispot).

SECONDARY OUTCOMES:
To develop test procedures in order to evaluate humoral and cellular anti-Tat immunity for future efficacy trials.

CONTACTS AND LOCATIONS:
Overall Officials: Pasquale Narciso, MD, Principal Investigator — I.R.C.C.S. Spallanzani Hospital, Rome; Aldo Di Carlo, MD, Principal Investigator — S. Gallicano Hospital- Rome; Adriano Lazzarin, MD, Principal Investigator — San Raffaele Hospital - Milan
Locations (3):
- Italy (3):
  - San Raffaele Hospital, Milan
  - I.R.C.C.S. Spallanzani Hospital, Rome
  - Istituto Dermatologico S. Gallicano-IRCCS, Rome

REFERENCES:
- [Background] Ensoli B, Buonaguro L, Barillari G, Fiorelli V, Gendelman R, Morgan RA, Wingfield P, Gallo RC. Release, uptake, and effects of extracellular human immunodeficiency virus type 1 Tat protein on cell growth and viral transactivation. J Virol. 1993 Jan;67(1):277-87. doi: 10.1128/JVI.67.1.277-287.1993. PMID 8416373
- [Background] Ensoli B, Gendelman R, Markham P, Fiorelli V, Colombini S, Raffeld M, Cafaro A, Chang HK, Brady JN, Gallo RC. Synergy between basic fibroblast growth factor and HIV-1 Tat protein in induction of Kaposi's sarcoma. Nature. 1994 Oct 20;371(6499):674-80. doi: 10.1038/371674a0. PMID 7935812
- [Background] Ensoli B, Barillari G, Salahuddin SZ, Gallo RC, Wong-Staal F. Tat protein of HIV-1 stimulates growth of cells derived from Kaposi's sarcoma lesions of AIDS patients. Nature. 1990 May 3;345(6270):84-6. doi: 10.1038/345084a0. PMID 2184372
- [Background] Ensoli B, Fiorelli V, Ensoli F, Cafaro A, Titti F, Butto S, Monini P, Magnani M, Caputo A, Garaci E. Candidate HIV-1 Tat vaccine development: from basic science to clinical trials. AIDS. 2006 Nov 28;20(18):2245-61. doi: 10.1097/QAD.0b013e3280112cd1. No abstract available. PMID 17117011
- See also: Related Info — http://www.hiv1tat-vaccines.info